CLINICAL TRIAL: NCT03906539
Title: Effect of Virgin Coconut Oil (VCO) on Cardiometabolic Parameters in Patients With Dyslipidemia: A Randomized, add-on, Placebo-controlled Clinical Trial
Brief Title: Effect of Virgin Coconut Oil (VCO) on Cardiometabolic Parameters in Patients With Dyslipidemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Collaborators: Coconut Development Board, Government of India (Unknown)
Responsible Party: Principal Investigator, RITUPARNA MAITI, Additional Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T/EMF/Pharma/18/23
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Dyslipidemias
Keywords: Cardiometabolic parameters; Virgin coconut oil; Serum lipoprotein; Lipid peroxidation; Atorvastatin
MeSH Terms: conditions — Dyslipidemias | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): The patients in control groups will receive tablet atorvastatin (10 mg/day) and a placebo capsule.
  Interventions: Drug: Atorvastatin 10mg; Other: Placebo
- VCO Group (Experimental): The VCO group will receive capsule VCO (1000mg/day) as an add-on to tablet atorvastatin (10 mg/day).
  Interventions: Drug: Atorvastatin 10mg; Dietary Supplement: Virgin Coconut Oil (VCO)

INTERVENTIONS:
Drug: Atorvastatin 10mg — Atorvastatin 10 mg per day
Dietary Supplement: Virgin Coconut Oil (VCO) — Capsule VCO (1000 mg/day)
  Arms: VCO Group
Other: Placebo — Placebo capsule - 1 capsule per day
  Arms: Control Group

SUMMARY:
The present research will help to assess the effect of virgin coconut oil on cholesterol level and also will help to know whether virgin coconut oil can reduce the risk of heart diseases or not.

DETAILED DESCRIPTION:
Dyslipidemia is a well-established risk factor for cardiovascular (CV) diseases. Lipid abnormalities, including high levels of low-density lipoprotein cholesterol (LDL-C), elevated triglycerides and low levels of high-density lipoprotein cholesterol (HDL-C), are independent predictors of CV disease. The National Cholesterol Education Program Adult Treatment Panel III (ATP III) guideline and the American College of Cardiology (ACC) and American Heart Association (AHA) guideline recommend the use of statins for primary prevention based on a patient's cardiovascular risk profile and low-density lipoprotein cholesterol (LDL-C) level. However, statin therapy may be insufficient for patients with mixed dyslipidemia, especially those with metabolic syndromes. While the addition of niacin, fibrate or ezetimibe may be useful in this setting, the combination therapy may lead to more adverse drug reactions.

Virgin Coconut Oil (VCO), a nutraceutical, is an oil obtained from the fresh, mature kernel of the coconut by mechanical or natural means, with or without the use of heat and without undergoing chemical refining and it contains a considerable amount of medium-chain fatty acids similar to those in mother's milk. The beneficial effects of VCO in the reduction of cardiovascular risk have been proved from previous animal and clinical studies. The previous study demonstrated the potential beneficiary effect of VCO in lowering lipid levels in serum and LDL oxidation by physiological oxidants and this property of VCO was attributed to the biologically active polyphenol components present in the oil. It has been also demonstrated the hypolipidemic effect of VCO through activation of lipoprotein lipase, lecithin cholesterol acyltransferase and enhanced formation of bile acids. It was found that isolated polyphenols from VCO can prevent cadmium-induced lipid abnormalities and cardiovascular risk ratios by improving antioxidant defence systems. VCO may improve cardiovascular and hepatic complications in obesity. The findings from another study suggest a beneficial eﬀect of VCO on lipid profile, renal status, hepatic antioxidant defence system, and cardiovascular risk indices in rats. It has been observed that VCO increased HDL-C level in patients with coronary artery disease (CAD). In a randomized crossover trial, it was found that daily consumption of VCO in young healthy adults significantly increased high-density lipoprotein cholesterol without any safety issues.

Our literature search revealed that to date, no clinical trial evaluated the potential of VCO as an add-on hypolipidemic agent in patients suffering from dyslipidemia. So, the present clinical trial has been designed to evaluate the effect of VCO on cardiometabolic parameters as an add-on with statins in patients with dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dyslipidemia [diagnosis of dyslipidemia is made when either of the lipid abnormality is present: LDL-C >140mg/dl, HDL-C <40mg/dl, Triglyceride >150mg/dl according to diagnostic criteria of dyslipidemia ]
* Patients aged 18-65 years, of either sex.
* Treatment-naive patients or patients who had not taken any treatment for at least 2 weeks before inclusion.

Exclusion Criteria:

* History of any cardiovascular diseases, stroke, diabetes, malignancy, musculoskeletal or hepatic diseases
* History of hypersensitivity to statins or coconut oil
* Patients who are already under treatment for the presenting conditions.
* Patients with drug/alcohol abuse.
* Pregnant and nursing women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in serum High Density Lipoprotein (HDL) | Baseline and 8 weeks
  Will be measured by autoanalyser

SECONDARY OUTCOMES:
Change in serum Lipoprotein (a) | Baseline and 8 weeks
  Will be measured by ELISA
Change in Atherogenic index | Baseline and 8 weeks
  Ratio of LDL cholesterol and HDL cholesterol
Change in Coronary risk index | Baseline and 8 weeks
  Ratio of total cholesterol and HDL cholesterol
Change in Cardiovascular risk index | Baseline and 8 weeks
  Ratio of triglyceride and HDL cholesterol
Change in visceral fat | Baseline and 8 weeks
  Will be analysed by by digital body fat analyser
Change in lipid peroxidation | Baseline and 8 weeks
  Thiobarbituric acid reactive substances (TBARS) will be estimated by spectrofluorometric method
Change in serum Low Density Lipoprotein (LDL) | Baseline and 8 weeks
  Will be measured by autoanalyser
Change in serum Very Low Density Lipoprotein (VLDL) | Baseline and 8 weeks
  Will be measured by autoanalyser
Change in serum total cholesterol | Baseline and 8 weeks
  Will be measured by autoanalyser
Change in serum triglyceride | Baseline and 8 weeks
  Will be measured by autoanalyser

CONTACTS AND LOCATIONS:
Locations (1):
- AIIMS, Bhubaneswar, Bhubaneshwar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yusuf S, Hawken S, Ounpuu S, Dans T, Avezum A, Lanas F, McQueen M, Budaj A, Pais P, Varigos J, Lisheng L; INTERHEART Study Investigators. Effect of potentially modifiable risk factors associated with myocardial infarction in 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):937-52. doi: 10.1016/S0140-6736(04)17018-9. PMID 15364185
- [Result] Gordon DJ, Probstfield JL, Garrison RJ, Neaton JD, Castelli WP, Knoke JD, Jacobs DR Jr, Bangdiwala S, Tyroler HA. High-density lipoprotein cholesterol and cardiovascular disease. Four prospective American studies. Circulation. 1989 Jan;79(1):8-15. doi: 10.1161/01.cir.79.1.8. PMID 2642759
- [Result] Sarwar N, Danesh J, Eiriksdottir G, Sigurdsson G, Wareham N, Bingham S, Boekholdt SM, Khaw KT, Gudnason V. Triglycerides and the risk of coronary heart disease: 10,158 incident cases among 262,525 participants in 29 Western prospective studies. Circulation. 2007 Jan 30;115(4):450-8. doi: 10.1161/CIRCULATIONAHA.106.637793. Epub 2006 Dec 26. PMID 17190864
- [Result] Bansal S, Buring JE, Rifai N, Mora S, Sacks FM, Ridker PM. Fasting compared with nonfasting triglycerides and risk of cardiovascular events in women. JAMA. 2007 Jul 18;298(3):309-16. doi: 10.1001/jama.298.3.309. PMID 17635891
- [Result] Grundy SM, Cleeman JI, Merz CN, Brewer HB Jr, Clark LT, Hunninghake DB, Pasternak RC, Smith SC Jr, Stone NJ; National Heart, Lung, and Blood Institute; American College of Cardiology Foundation; American Heart Association. Implications of recent clinical trials for the National Cholesterol Education Program Adult Treatment Panel III guidelines. Circulation. 2004 Jul 13;110(2):227-39. doi: 10.1161/01.CIR.0000133317.49796.0E. PMID 15249516
- [Result] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW, Eddleman KM, Jarrett NM, LaBresh K, Nevo L, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S1-45. doi: 10.1161/01.cir.0000437738.63853.7a. Epub 2013 Nov 12. No abstract available. PMID 24222016
- [Result] Famurewa AC, Ekeleme-Egedigwe CA, Nwali SC, Agbo NN, Obi JN, Ezechukwu GC. Dietary Supplementation with Virgin Coconut Oil Improves Lipid Profile and Hepatic Antioxidant Status and Has Potential Benefits on Cardiovascular Risk Indices in Normal Rats. J Diet Suppl. 2018 May 4;15(3):330-342. doi: 10.1080/19390211.2017.1346031. Epub 2017 Aug 17. PMID 28816548
- [Result] Nevin KG, Rajamohan T. Beneficial effects of virgin coconut oil on lipid parameters and in vitro LDL oxidation. Clin Biochem. 2004 Sep;37(9):830-5. doi: 10.1016/j.clinbiochem.2004.04.010. PMID 15329324
- [Result] Arunima S, Rajamohan T. Virgin coconut oil improves hepatic lipid metabolism in rats--compared with copra oil, olive oil and sunflower oil. Indian J Exp Biol. 2012 Nov;50(11):802-9. PMID 23305031
- [Result] [Should the specialist examination be introduced? Thoughts of the Education Committee]. Ugeskr Laeger. 1969 Jan 23;131(4):170-1. No abstract available. Danish. PMID 5787998
- [Result] Panchal SK, Carnahan S, Brown L. Coconut Products Improve Signs of Diet-Induced Metabolic Syndrome in Rats. Plant Foods Hum Nutr. 2017 Dec;72(4):418-424. doi: 10.1007/s11130-017-0643-0. PMID 29079969
- [Result] Cardoso DA, Moreira AS, de Oliveira GM, Raggio Luiz R, Rosa G. A COCONUT EXTRA VIRGIN OIL-RICH DIET INCREASES HDL CHOLESTEROL AND DECREASES WAIST CIRCUMFERENCE AND BODY MASS IN CORONARY ARTERY DISEASE PATIENTS. Nutr Hosp. 2015 Nov 1;32(5):2144-52. doi: 10.3305/nh.2015.32.5.9642. PMID 26545671
- [Result] Chinwong S, Chinwong D, Mangklabruks A. Daily Consumption of Virgin Coconut Oil Increases High-Density Lipoprotein Cholesterol Levels in Healthy Volunteers: A Randomized Crossover Trial. Evid Based Complement Alternat Med. 2017;2017:7251562. doi: 10.1155/2017/7251562. Epub 2017 Dec 14. PMID 29387131
- [Result] Teramoto T, Sasaki J, Ueshima H, Egusa G, Kinoshita M, Shimamoto K, Daida H, Biro S, Hirobe K, Funahashi T, Yokote K, Yokode M; Japan Atherosclerosis Society (JAS) Committee for Epidemiology and Clinical Management of Atherosclerosis. Diagnostic criteria for dyslipidemia. Executive summary of Japan Atherosclerosis Society (JAS) guideline for diagnosis and prevention of atherosclerotic cardiovascular diseases for Japanese. J Atheroscler Thromb. 2007 Aug;14(4):155-8. doi: 10.5551/jat.e537. No abstract available. PMID 17827859
- [Result] Ermakova GL, Abakumov EM, Martynova VA. [Immunological and microbiological parallels in pneumonia complicating leukemia]. Klin Med (Mosk). 1973 Feb;51(2):29-32. No abstract available. Russian. PMID 4700825